CLINICAL TRIAL: NCT02327559
Title: Randomized Controlled Trial of a Mindfulness Intervention for Labor-Related Pain and Fear
Brief Title: Prenatal Education About Reducing Labor Stress (PEARLS)
Acronym: PEARLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Mount Zion Health Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PEARLSMZHF
Record Dates: First submitted 2014-06-23; First posted 2014-12-30 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Labor Pain; Tocophobia
Keywords: childbirth; mindfulness; fear of labor; labor pain; coping; self-efficacy; childbirth satisfaction; depression
MeSH Terms: conditions — Labor Pain; Depression | interventions — Parturition; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mind in Labor (MIL) (Experimental): Mind in Labor: Working with Pain in Childbirth (MIL) is a 16-hour mindfulness-based childbirth education course. It is an abbreviated weekend workshop form of the 9-week Mindfulness-Based Childbirth and Parenting (MBCP) education program, which is a tailored form of Mindfulness-Based Stress Reduction.
  Interventions: Behavioral: Mind in Labor (MIL): Working with Pain in Childbirth
- Treatment As Usual (TAU) (Active Comparator): Treatment As Usual (TAU) refers to standard hospital- and community-based childbirth preparation courses (high quality childbirth education that excludes a mindfulness or mind/body stress reduction focus).
  Interventions: Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Mind in Labor (MIL): Working with Pain in Childbirth — The Mind in Labor (MIL) mindfulness intervention for pregnant women and their partners integrates mindfulness strategies for coping with labor pain and fear and formal mindfulness meditation with traditional childbirth education. The MIL intervention is held over 3 consecutive weekend days (Friday - Sunday) for a total of 16 hours of mindfulness skills training for childbirth preparation and labor pain management. Mindfulness strategies for coping with labor-related pain and fear are taught in an interactive, experiential format, with periods of didactic instruction.
  Arms: Mind in Labor (MIL)
Behavioral: Treatment as usual (TAU) — The treatment as usual "TAU" active comparison condition includes participation in a standard care childbirth education course, chosen by participants in the TAU arm from a pre-approved list of hospital- and community-based childbirth education courses comparable in length and quality to MIL, but without any mindfulness meditation, mindful movement/yoga, or other core mind/body component (e.g., hypnosis).
  Arms: Treatment As Usual (TAU)

SUMMARY:
The purpose of this small randomized controlled trial (RCT) is to compare the impact of a brief (16 hour) 3rd trimester mindfulness-based childbirth education program, "Mind in Labor (MIL): Working with Pain in Childbirth," with a standard care/"treatment as usual" (TAU) active control condition of standard hospital- and community-based childbirth education. The MIL group is expected to demonstrate a reduction in fear of labor (less pain catastrophizing and greater childbirth self-efficacy), less perceived pain in labor, less use of pain medication in labor, greater birth satisfaction, and better prenatal and postpartum psychological adjustment compared to the TAU group.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* No prior full-term pregnancy or live birth prior to the current pregnancy
* In 3rd trimester of healthy, singleton pregnancy
* Willingness to be randomized
* Able to read, write, and understand spoken English
* Planned hospital birth in the San Francisco Bay Area

Exclusion Criteria:

* Current or prior formal meditation experience
* Formal yoga practice prior to pregnancy (brief prenatal yoga practice will not lead to exclusion)
* Participation in other mind/body childbirth preparation course (e.g., with hypnosis focus)
* Planned elective Cesarean birth
* Planned homebirth or other non-hospital birth setting

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-10; Primary Completion 2014-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in Fear of labor (childbirth self-efficacy and pain catastrophizing) | Baseline (pre-intervention, 3rd trimester); Post-intervention (prior to birth)
  Change in levels of self-reported childbirth self-efficacy and pain catastrophizing
Perceived labor pain | Postpartum (average of 6 weeks post-birth)
  Retrospective self-report of perceived pain in labor
Pain medication use during labor | Labor (during childbirth)
  Type, dose, and frequency of pain medication use during labor and delivery, recorded in medical record.
Childbirth satisfaction | Postpartum (average of 6 weeks post-birth)
  Self-reported satisfaction with experiences of childbirth
Change in Depression | Baseline (pre-intervention, 3rd trimester); Post-intervention (prior to birth); Postpartum (average of 6 weeks postbirth); Follow-up (1-2 years post-birth)
  Self-reported depressive mood/symptoms of depression

SECONDARY OUTCOMES:
Perceived stress and parenting stress | Baseline (pre-intervention, 3rd trimester); Post-intervention (prior to birth); Postpartum (average of 6 weeks postbirth); Follow-up (1-2 years post-birth)
  Change in and level of self-report of general perceived life stress and parenting-specific stress
Mindfulness and interoceptive body awareness | Baseline (pre-intervention, 3rd trimester); Post-intervention (prior to birth); Postpartum (average of 6 weeks postbirth); Follow-up (1-2 years post-birth)
  Change in and level of self-report mindfulness in everyday life and interoceptive body awareness
Positive and negative emotion | Baseline (pre-intervention, 3rd trimester); Post-intervention (prior to birth); Postpartum (average of 6 weeks postbirth); Follow-up (1-2 years post-birth)
  Change in and level of self-report of intensity and frequency of positive and negative affect
Anxiety | Baseline (pre-intervention, 3rd trimester); Post-intervention (prior to birth); Postpartum (average of 6 weeks postbirth); Follow-up (1-2 years post-birth)
  Change in and level of self-report of trait anxiety, pregnancy-related anxiety, and worry

CONTACTS AND LOCATIONS:
Overall Officials: Larissa G Duncan, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- The Osher Center for Integrative Medicine, San Francisco, California, United States

REFERENCES:
- [Derived] O'Connell MA, Khashan AS, Leahy-Warren P, Stewart F, O'Neill SM. Interventions for fear of childbirth including tocophobia. Cochrane Database Syst Rev. 2021 Jul 7;7(7):CD013321. doi: 10.1002/14651858.CD013321.pub2. PMID 34231203
- [Derived] Sbrilli MD, Duncan LG, Laurent HK. Effects of prenatal mindfulness-based childbirth education on child-bearers' trajectories of distress: a randomized control trial. BMC Pregnancy Childbirth. 2020 Oct 15;20(1):623. doi: 10.1186/s12884-020-03318-8. PMID 33059638
- [Derived] Duncan LG, Cohn MA, Chao MT, Cook JG, Riccobono J, Bardacke N. Benefits of preparing for childbirth with mindfulness training: a randomized controlled trial with active comparison. BMC Pregnancy Childbirth. 2017 May 12;17(1):140. doi: 10.1186/s12884-017-1319-3. PMID 28499376